CLINICAL TRIAL: NCT00149734
Title: Atypical Antipsychotics and P50 Sensory Gating
Brief Title: Addition of Ondansetron to Ongoing Antipsychotic Treatment for Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-0255; R01MH050787 (NIH); COMIRB # 04-0255; DNBBS 73-MCR
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Ondansetron; P50 sensory gating; Evoked potentials; 5-HT3 receptors; Atypical antipsychotics
MeSH Terms: conditions — Schizophrenia | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron followed by placebo (Experimental): Participants will take ondansetron then placebo plus an atypical antipsychotic drug
  Interventions: Drug: Ondansetron followed by placebo
- Placebo followed by Ondansetron (Experimental): Participants will take placebo then ondansetron plus an atypical antipsychotic drug
  Interventions: Drug: Placebo followed by Ondansetron

INTERVENTIONS:
Drug: Ondansetron followed by placebo — Participants will take 16mg of ondansetron daily for the first three months followed by 3 months of placebo. An atypical antipsychotic drug (olanzapine,quetiapine, or aripiprazole) will also be taken throughout the 6 months treatment period.
  Other Names: Zofran, Zuplenz
  Arms: Ondansetron followed by placebo
Drug: Placebo followed by Ondansetron — Participants will take placebo daily for the first three months followed by 3 months of 16mg of ondansetron daily. An atypical antipsychotic drug (olanzapine,quetiapine, or aripiprazole) will also be taken throughout the 6 months treatment period.
  Other Names: Zofran, Zuplenz
  Arms: Placebo followed by Ondansetron

SUMMARY:
This study will examine the effects of ondansetron on auditory nerve activity in people with schizophrenia who are being treated with new antipsychotics.

DETAILED DESCRIPTION:
Schizophrenia is a devastating brain disorder. Most people with schizophrenia have difficulty filtering out unimportant auditory information. They have an inability to appropriately inhibit, or gate, sensory information that enters the ear. Standard treatments do not address this problem. When the drug ondansetron is taken in addition to typical antipsychotic drugs, P50 auditory gating improves. However, ondansetron has not been used with some of the newer, atypical antipsychotic drugs. This study will evaluate the effect of combining ondansetron with newer, atypical antipsychotic drugs on P50 auditory gating.

Participants in this double-blind study will be randomly assigned to receive either ondansetron or placebo for 3 months. Upon completion of the first 3 months, participants will be crossed over to receive the other treatment for an additional 3 months. All participants will also take an atypical antipsychotic drug, including olanzapine, quetiapine, or aripiprazole. Auditory gating will be assessed using computerized cognitive testing and functional magnetic resonance imaging (fMRI) at baseline and Months 3 and 6. Vital signs and evoked potentials will be assessed at Weeks 1, 3, and 6. Clinical symptoms and cognitive abilities will also be evaluated to determine the effectiveness of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia
* Stable, chronic schizophrenia
* Currently taking atypical medications
* Use of effective form of contraception throughout study

Exclusion Criteria:

* History of any alcohol or drug abuse within 3 months of study start date
* Any other major neurological disorders
* History of or current head trauma
* Any medical conditions affecting the central nervous system
* Current epilepsy, asthma, migraine headache, previous myocardial infarction, stroke, diabetes, hypertension, narrow angle glaucoma, or neuromuscular illnesses
* Pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence E. Adler, MD, Principal Investigator — University of Colorado Health Sciences Center, VISN19 MIRECC
Locations (1):
- Denver VAMC, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler LE, Cawthra EM, Donovan KA, Harris JG, Nagamoto HT, Olincy A, Waldo MC. Improved p50 auditory gating with ondansetron in medicated schizophrenia patients. Am J Psychiatry. 2005 Feb;162(2):386-8. doi: 10.1176/appi.ajp.162.2.386. PMID 15677607
- [Background] Adler LE, Olincy A, Cawthra EM, McRae KA, Harris JG, Nagamoto HT, Waldo MC, Hall MH, Bowles A, Woodward L, Ross RG, Freedman R. Varied effects of atypical neuroleptics on P50 auditory gating in schizophrenia patients. Am J Psychiatry. 2004 Oct;161(10):1822-8. doi: 10.1176/ajp.161.10.1822. PMID 15465979

RESULTS

PARTICIPANT FLOW:
Groups:
- Ondansetron Followed by Placebo: Participants will take ondansetron (16mg) at one study visit, then a placebo at another study visit one week later.
- Placebo Followed by Ondansetron: Participants will take a placebo at one study visit, then ondansetron (16mg) at another study visit one week later.
Period: Overall Study
Arm/Group | Ondansetron Followed by Placebo | Placebo Followed by Ondansetron
Started | 4 | 4
Started Intervention 2 | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No information is available regarding the demographics within separate arms/groups. Multiple attempts were made to obtain results information. However, the PI has retired and the only data available is for all participants.
Groups:
- All Participants: Ondansetron followed by placebo group and Placebo followed by Ondansetron group
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: P50 Sensory Gating
Description: P50 Sensory Gating as measured by evoked potentials (response to stimuli, in this case, clicking sounds).The P50 potential was identified and measured using a computer algorithm. The amplitude of the P50 test wave was divided by the amplitude of the P50 conditioning wave, expressed as a percentage: the P50 ratio. Lower P50 ratios represent better outcomes.
Time Frame: Up to 3 hours
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Ondansetron: Ondansetron (16 mg)
- Placebo: Placebo
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 8 | 8
percentage | 41.4 (39.7) | 80.2 (21.3)

2. Primary Outcome: Cognitive Testing
Time Frame: Measured at Months 3 and 6
Population: this outcome measure was not collected due to a change in the study design via a protocol amendment.
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No adverse events data is available. The PI has left the university and has confirmed that he no longer has access to the data, and the remaining members of the study team confirmed that the data no longer exists. Therefore, the number of participants "At risk" is 0, because no participants could be analyzed for adverse events.
Arm/Group | Ondansetron | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limited data is available. The PI has left the university and has confirmed that he no longer has access to the data, and the remaining members of the study team confirmed that the data no longer exists.

The study design was altered after registration due to a protocol amendment to not do a long-term study but to directly study participants on long-term clozapine treatment (a 5HT3 receptor antagonist like ondansetron) with other antipsychotics, including atypicals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No